CLINICAL TRIAL: NCT05481021
Title: Assessing the Frequency of Burnout Syndrome Among Diabetes Specialist Trainee Registrars in United Kingdom and Identifying Any Associated Factors
Brief Title: Burnout Syndrome Among Diabetes Specialist Trainee Registrars in United Kingdom
Status: Completed | Type: Observational
Sponsor: United Arab Emirates University (Other)
Responsible Party: Principal Investigator, Dr Adnan Agha, Assistant Professor, Internal Medicine, College of Medicine and Health Sciences, United Arab Emirates University, United Arab Emirates University
Other Study IDs: UAEU_CMHS_IM_ERSC_2022_1166
Record Dates: First submitted 2022-07-27; First posted 2022-07-29 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Burnout, Professional; Work-Related Condition
Keywords: Burnout syndrome; Diabetes; Specialist trainee Registrar; Physician burnout; United Kingdom
MeSH Terms: conditions — Burnout, Professional; Burnout, Psychological; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Diabetes Specialist trainee Registrars/Middle grade working in UK: All doctors in in middle grade or similar rank who are in training as Diabetes Specialist trainee Registrars or non-trainee Middle grade doctors working in Diabetes/Endocrinology department in NHS Wales, NHS Scotland or Health and Social Care northern Ireland (health systems in all of UK)
  Interventions: Other: No intervention but assessing for burnout syndrome in all group

INTERVENTIONS:
Other: No intervention but assessing for burnout syndrome in all group — Using Maslach Burnout inventory to assess the presence of burnout and a self reporting questionnaire to identify possible stressors or associations

SUMMARY:
Burnout Syndrome is a medical condition caused by long-term job-related strain and is defined by presence of either one or more of the three states i.e. emotional exhaustion, depersonalization and lack of personal accomplishment. Burnout has been shown to cause decreased work output and mental well being of employees and increase errors at workplace. Burnout is observed in various lines of work and but has been found to be especially high among healthcare professionals. Diabetes Mellitus is a generally a life-long condition and diabetes specialists deal with patients of this chronic condition frequently. The burnout among diabetes specialist trainees in United Kingdom was found to be over 50% in a study done in pre-pandemic times in 2018 and there is a need to repeat this study to see if there any change in terms of presence of burnout in this group of health care professionals.

DETAILED DESCRIPTION:
Burnout syndrome can develop after a prolonged response to chronic emotional and interpersonal workplace stressors, and is defined by 3 dimensions - emotional exhaustion, depersonalization and lack of personal accomplishment. The consequences of burnout on an employee can be on a psychological and somatic level as well as on her/his ability to perform work, and hospital physicians with burnout have higher sickness and absenteeism and decreases work output. Burnout among physicians can also lead to medical mistakes and increasing the odds for workplace failure with adverse affects in their attitude towards their work. Research has shown that doctors reporting high workload and a unsupported work climate have higher stress, burnout and dissatisfaction with their career.

Study done by author previously in 2018 among Diabetes specialist registrars in England Scotland and Wales identified burnout syndrome in 57.5% respondents with commonest self-reported stressors being workload and lack of specialty training. In order to address this problem nationally, there is need to re-assess the presence of burnout and then consider planning for any interventional steps that may help reduce burnout.

ELIGIBILITY:
Inclusion Criteria:

1. All specialty doctors working in Diabetes or Endocrinology department post foundation years, in the following deaneries/regions in United Kingdom

   * Health Education Yorkshire & Humber
   * Health Education East Midlands
   * Health Education East of England
   * Health Education Kent Surrey & Sussex
   * Health Education North West & Mersey Deanery
   * Health Education North East
   * Health Education South West Peninsula and Severn Deanery
   * Health Education Thames Valley (Oxford)
   * Health Education Wessex
   * Health Education West Midlands
   * London Deanery (North West, North Central & East London, South London)
   * Northern Ireland Medical & Dental Training Agency
   * Scotland Deanery (West, South East, East, North)
   * Wales Deanery
2. Doctors currently working for the last 3 months in either one of the following posts:

   * Clinical fellow/ non-deanery training post/locally employed trainee
   * Academic clinical fellow trainee / ACF
   * Core Trainee or Specialist trainee year 3/ awaiting National Training Number
   * Associate Specialist Equivalent/Trust middle grade
   * Specialist trainee year 4 through year 8
   * Clinical Lecturer
   * Diabetes consultant (new i.e within 3 years of appointment, locum, fixed term or substantive)
3. Currently working in UK for at least six months in the last one year
4. Agreeing to participate via informed consent

Exclusion Criteria:

* Self-reported presence of mental health illness and/or active treatment.
* Not currently working for more than 3 months e.g on sick leave.

Ages: 21 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: All the doctors fulfilling the above criteria will be sent an online invite to participate in this survey via national organizations on their emails as well as via official online platform. The online forms will remain open over 3 months period. The participants meeting the above-mentioned criteria will be selected and they will complete the self-reported profroma containing demographics and Maslach burnout inventory ( a validated tool via Mind Garden TM for Burnout Syndrome) on an online secure platform. No personal identifiable information will be collected or stored and the results will be displayed in the form of deanery / national cumulative results.
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2022-07-05 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Identify burnout | 6 months
  To assess the frequency of burnout syndrome in Diabetes and Endocrinology specialty trainee registrars in all of United Kingdom by using a validated tool via Mind Garden, Malasch Inventory for Burnout Syndrome, latest edition 2016, assessing all three subscales of burnout i.e Emotional Exhaustion (with cutoff score for high burnout as per standardized z value = Mean + (SD* 0.5); range 0-54 with higher scores meaning a worse outcome), Depersonalization (with cutoff score for high burnout as per standardized z value = Mean + (SD * 1.25); range 0-30 with higher scores meaning a worse outcome), and lack of personal accomplishment (with cutoff score for high burnout per standardized z value = Mean + (SD * 0.10); range 0-48 with higher scores meaning a better outcome)
Identify any self-reported stressors associated with burnout | 6 months
  To assess the presence of associated self-reported factors for burnout syndrome

SECONDARY OUTCOMES:
To compare any change in presence of burnout from previous cross-sectional study (5 years ago) | 12 months
  To compare the frequency of burnout syndrome in Diabetes and Endocrinology specialty trainee registrars in all of UK done in 2022-2023 with frequency of burnout syndrome in Diabetes and Endocrinology specialty trainee registrars in 2018 (previous survey published and data available for comparison.

CONTACTS AND LOCATIONS:
Overall Officials: Adnan Agha, Principal Investigator — United Arab Emirates University, College of Medicine & Health Sciences
Locations (1):
- Internal Medicine, College of Medicine and Health Sciences, Al Ain City, Abu Dhabi Emirate, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Undecided
The individual data will be non identifiable and without personal identifiable information. can consider collaboration with other researchers at later stage

REFERENCES:
- [Background] Agha A, Basu A, Hanif W. Burnout in diabetes and endocrinology specialist registrars across England, Scotland and Wales in the pre-COVID era. Prim Care Diabetes. 2022 Aug;16(4):515-518. doi: 10.1016/j.pcd.2022.05.005. Epub 2022 Jun 3. PMID 35667990
- [Background] Gundersen L. Physician burnout. Ann Intern Med. 2001 Jul 17;135(2):145-8. doi: 10.7326/0003-4819-135-2-200107170-00023. No abstract available. PMID 11453722
- [Background] Agha A, Mordy A, Anwar E, Saleh N, Rashid I, Saeed M. Burnout among middle-grade doctors of tertiary care hospital in Saudi Arabia. Work. 2015;51(4):839-47. doi: 10.3233/WOR-141898. PMID 24962300
- [Derived] Agha A, Basu A, Anwar E, Hanif W. Burnout among diabetes specialist registrars across the United Kingdom in the post-pandemic era. Front Med (Lausanne). 2024 Mar 26;11:1367103. doi: 10.3389/fmed.2024.1367103. eCollection 2024. PMID 38596789
- See also: The gold standard for burnout assessment. Maslach Burnout Inventory — http://www.mindgarden.com/117-maslach-burnout-inventory-mbi